CLINICAL TRIAL: NCT03062566
Title: Prognostic Potential of Prehospital S100B, Glial Fibrillary Acidic Protein (GFAP) and Neuron Specific Annuals (NSE) Levels in Patients Suffering Severe Traumatic Brain Injury (TBI)
Brief Title: Prognostic Potential of Prehospital Biomarkers in TBI Patients
Acronym: PreTBI III
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Protokol_v3_240816_PreTBI_III
Record Dates: First submitted 2016-11-21; First posted 2017-02-23 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2018-05

CONDITIONS: Traumatic Brain INjury
Keywords: biomarkers; point-of-care analysis
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Severe TBI patients: GCS 3-8
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling from peripheral venous catheter routinely inserted in trauma patients during transportation

SUMMARY:
The PreTBI III study aims to investigate the prognostic potential of prehospital and repeated in-hospital S100B, NSE and GFAP measurements as predictors of neurological outcome in patients suffering severe TBI. Knowledge on prehospital S100B, GFAP and NSE levels as predictors of neurological outcome and mortality may underline the potential of a point-of-care analysis. Possibly, the early biomarker levels may contributed to accurate monitoring of biomarker dynamics and hereby support neurosurgeons and anaesthetists in the clinical decision-making regarding treatment and level of care offered to the patient.

Hypotheses:

1. Prehospital S100B level is a significant predictor of unfavourable neurological outcome (dichotomized disability rating scale (DRS) and glasgow outcome scale extended (GOS-E) measures) in severe TBI patients.
2. Prehospital GFAP level is a significant predictor of unfavourable neurological outcome (dichotomized DRS and GOSE measures) in severe TBI patients.
3. Prehospital NSE level is a significant predictor of unfavourable neurological outcome (dichotomized DRS and GOSE measures) in severe TBI patients.
4. combined panel of prehospital S100B, GFAP and NSE levels is a significant predictor of unfavourable neurological outcome (dichotomized DRS and GOSE measures) in severe TBI patients.
5. Unfavourable neurological outcome (dichotomized DRS and GOSE measures) in severe TBI patients can be predicted by dynamics in repeated measurements of S100B, GFAP and NSE.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with Glasgow Coma Score (GCS) GCS 3-8 suffering relevant trauma and displaying relevant clinical indices compatible with TBI as evaluated by EMS staff. Patients are considered incompetent due to on-going alteration of mental state.

Exclusion Criteria:

* >6 hours elapsed after trauma, unknown time of trauma, multi trauma, known dementia, chronic psychosis or active central nervous system (CNS) pathology.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years) suffering isolated head trauma and receiving an ambulance dispatched by the Prehospital Emergency Medical Services (EMS) in the Central Denmark Region.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of se-S100B in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Specificity of se-S100B in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Positive predictive value of se-S100B in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Negative predictive value of se-S100B in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)

SECONDARY OUTCOMES:
Sensitivity of se-GFAP in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Specificity of se-GFAP in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Positive predictive value of se-GFAP in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Negative predictive value of se-GFAP in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Sensitivity of se-NSE in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Specificity of se-NSE in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Positive predictive value of se-NSE in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Negative predictive value of se-NSE in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)

OTHER OUTCOMES:
Mortality rates corresponding to se-S100B values | in relation to event within 1 year of trauma
  survival versus death <7 days, 3 months and 6 months after trauma 6-month
Mortality rates corresponding to se-GFAP values | in relation to event within 1 year of trauma
  survival versus death <7 days, 3 months and 6 months after trauma 6-month
Mortality rates corresponding to se-NSE values | in relation to event within 1 year of trauma
  survival versus death <7 days, 3 months and 6 months after trauma 6-month
Sensitivity of combined se-S100B, se-GFAP and se-NSE in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
Specificity of combined se-S100B, se-GFAP and se-NSE in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
Positive predictive value of combined se-S100B, se-GFAP and se-NSE in relation to a binary outcome measured by by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
Negative predictive value of combined se-S100B, se-GFAP and se-NSE in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
Biomarker dynamics between prehospital and in-hospital se-S100B values in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
Biomarker dynamics between prehospital and in-hospital se-GFAP values in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
Biomarker dynamics between prehospital and in-hospital se-NSE values in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
Biomarker dynamics between prehospital and in-hospital combination of se-S100B, se-GFAP and se-NSE values in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital Emergency Medical Services, Central Denmark Region, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No